CLINICAL TRIAL: NCT03123484
Title: β-elemene Combine With EGFR-TKI for Advanced EGFR-TKI-resistant Non-Small Cell Lung Cancer
Brief Title: β-elemene Combine With EGFR-TKI for Advanced EGFR-TKI-resistant NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University, China (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Liaoning Cancer Hospital & Institute (Other); Shengjing Hospital (Other); General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology,The First Hospital of China Medical University Affiliation: China Medical University, China, China Medical University, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOG1702
Record Dates: First submitted 2017-04-05; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: beta-elemene
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- β-elemene+EGFR TKI (Experimental): EGFR-TKIs(Erlotinib, Gefitinib and Icotinib) and β-elemene
  Interventions: Drug: β-elemene; Drug: EGFR-TKIs(Erlotinib, Gefitinib and Icotinib)
- EGFR TKI (Active Comparator): EGFR-TKIs(Erlotinib, Gefitinib and Icotinib)
  Interventions: Drug: EGFR-TKIs(Erlotinib, Gefitinib and Icotinib)

INTERVENTIONS:
Drug: β-elemene — β-elemene：400-600mg + 5%GS 500ml,ivgtt,qd, continuously 45days
  Other Names: elemene liposomes
  Arms: β-elemene+EGFR TKI
Drug: EGFR-TKIs(Erlotinib, Gefitinib and Icotinib) — EGFR-TKIs(Erlotinib, Gefitinib and Icotinib) as usual

SUMMARY:
Epidermal Growth Factor Receptor tyrosine-kinase inhibitors （EGFR-TKIs）, including gefitinib，erlotinib and icotinib demonstrate excellent effect on the treatment of non small cell lung cancer (NSCLC) patients with EGFR mutations. However, patients who are initially sensitive to the drugs eventually become resistance. In this study, the investigators aim to explore the efficacy of beta-elemene, combining with EGFR-TKI in advanced non-small cell lung cancer with EGFR-TKI resistance.

DETAILED DESCRIPTION:
Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs), including gefitinib，erlotinib and icotinib demonstrate excellent effect on the treatment of non-small cell lung cancer (NSCLC) patients with EGFR mutations. However, patients who are initially sensitive to the drugs eventually become resistance. Beta-elemene, a natural plant drug extracted from Curcuma wenyujin, has been used as an antitumor drug for different tumors, including NSCLC via mechanism that inhibits Ras/Mapk signaling and cell cycle progression.In this study, the investigators aim to explore the efficacy of beta-elemene, combining with EGFR-TKI in advanced non-small cell lung cancer with EGFR-TKI resistance.

main objectives: progression-free survival (PFS) ratio in 12 week the secondary goal: Objective Response Rate （ORR）

ELIGIBILITY:
Inclusion Criteria:

1. Obtain of informed consent.
2. Histologically or cytologically confirmed, inoperable, recurrence or metastasis advanced non-small cell lung cancer (TNM Stage ⅢB or stage Ⅳ), took EGFR-TKI longer than 6 months and appeared disease progression.
3. At least one measurable lesion (helical CT scan long diameter ≥10mm, meet the requirements of the standard Response Evaluation Criteria In Solid Tumors（RESCIST） version 1.1).
4. Eastern Cooperative Oncology Group（ECOG）Performance Status（PS） :0-2.
5. Aged from 18 to 75 years (18 and 75 years are included).
6. Life expectancy ≥12 weeks.
7. Adequate bone marrow reserve and organ function as follows:

   Absolute neutrophils count (ANC) ≥1.5 x 10 to the 9th power/L (band neutrophil and segmented neutrophil), platelets > 100 x 10 to the 9th power/L and Hb≥90g/L.

   Hepatic: total bilirubin less than or equal to 1.5 times upper limit of normal (ULN).

   Alkaline phosphatase (AP), alanine transaminase (ALT) and aspartate transaminase (AST) less than or equal to 3.0 times ULN (or less than or equal to 5 times ULN in case of known liver involvement.

   Renal: Serum Creatinine less than or equal to 1.25 times upper limit of normal (ULN).
8. Females of child-bearing potential must have negative serum pregnancy test. Sexually active males and females (of childbearing potential) willing to practice contraception during the study.

Exclusion Criteria:

1. Do not meet the above criteria.
2. Unhealed toxicity of prior anti-cancer treatment (CTCAE Level 1) or surgery.
3. Symptomatic Central Nervous System (CNS) metastases.
4. Clinical uncontrolled active infection, such as acute pneumonia, active hepatitis B or C (prior hepatitis B history, despite medication treatment control or not, HBV DNA≥500copies or ≥100IU/ml), etc.
5. Prior other malignant disease in 5 years (except carcinoma in situ of cervix, or non melanoma skin cancers, or localized prostate cancer with Gleason ≤6).
6. Take part in new drug clinical trials within one month or taking part in a trial now.
7. Pregnant or lactating woman.
8. Other conditions regimented at investigators' discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
PFS ratio in 12 week | 12 week
  progression free survival ratio in 12 week

SECONDARY OUTCOMES:
OR Rate | 12 week
  Objective Response Rate

CONTACTS AND LOCATIONS:
Overall Officials: Liu yunpeng, PhD, Principal Investigator — Director of Department of Medical Oncology,The First Hospital of China Medical University Affiliation: China Medical University, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xu XW, Yuan ZZ, Hu WH, Wang XK. [Meta-analysis on elemene injection combined with cisplatin chemotherapeutics in treatment of non-small cell lung cancer]. Zhongguo Zhong Yao Za Zhi. 2013 May;38(9):1430-7. Chinese. PMID 23944083
- [Background] Li QQ, Wang G, Huang F, Li JM, Cuff CF, Reed E. Sensitization of lung cancer cells to cisplatin by beta-elemene is mediated through blockade of cell cycle progression: antitumor efficacies of beta-elemene and its synthetic analogs. Med Oncol. 2013 Mar;30(1):488. doi: 10.1007/s12032-013-0488-9. Epub 2013 Feb 9. PMID 23397083
- [Background] Liu J, Hu XJ, Jin B, Qu XJ, Hou KZ, Liu YP. beta-Elemene induces apoptosis as well as protective autophagy in human non-small-cell lung cancer A549 cells. J Pharm Pharmacol. 2012 Jan;64(1):146-53. doi: 10.1111/j.2042-7158.2011.01371.x. Epub 2011 Oct 27. PMID 22150682
- [Background] Matsuoka H, Kaneda H, Sakai K, Koyama A, Nishio K, Nakagawa K. Clinical Response to Everolimus of EGFR-Mutation-Positive NSCLC With Primary Resistance to EGFR TKIs. Clin Lung Cancer. 2017 Jan;18(1):e85-e87. doi: 10.1016/j.cllc.2016.08.004. Epub 2016 Oct 4. No abstract available. PMID 28341110
- [Background] Passiglia F, Listi A, Castiglia M, Perez A, Rizzo S, Bazan V, Russo A. EGFR inhibition in NSCLC: New findings.... and opened questions? Crit Rev Oncol Hematol. 2017 Apr;112:126-135. doi: 10.1016/j.critrevonc.2017.02.009. Epub 2017 Feb 16. PMID 28325254